CLINICAL TRIAL: NCT03016429
Title: Safety and Clinical Outcomes of Magnetic Resonance Imaging in Patients With Cardiac Implantable Electrical Devices
Acronym: BIDMC-MRI
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Dan B. Kramer, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2016P000204
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cardiac Disease
Keywords: pacemaker; defibrillator; magnetic resonance imaging; cardiac implantable electronic device
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol outlines a prospective study evaluating safety and clinical outcomes of magnetic resonance imaging (MRI) examinations performed on patients with cardiac implantable electrical devices (CIEDs) including pacemakers (PMs) and implantable cardioverter-defibrillators (ICDs). This prospective study aims to improve the evidence base regarding this common clinical scenario. Specifically, the investigators aim to address whether results of MRI in PM/ICD patients affect physician decision making related to clinical management strategy and planning treatment interventions. Further, this study will evaluate whether the results of MRI in these patients affects patient outcomes related to survival and adverse events during or after MRI scanning.

DETAILED DESCRIPTION:
MRI is the preferred imaging modality for both acute and elective evaluation of many conditions. For example, for many diseases of the central nervous system, no other imaging modality provides the requisite soft tissue resolution to support critical care elements such as neurosurgical planning or assessment of intracranial malignancies.

Historically, MRIs were considered contraindicated for patients with CIEDs including PMs and ICDs. However, studies have demonstrated very high utilization of MRIs among patients eligible for CIEDs. In many cases, alternative imaging is either insufficient or, as with CT-myelography, poses substantial risks or procedural hurdles that may be less favorable than the potential risks of an MRI.

In recent years, a growing literature has suggested that MRIs can be performed safely in the setting of CIEDs if certain precautions are taken. Additionally, guidance documents have been released by professional societies including the American Heart Association (AHA) and the American College of Radiology (ACR) outlining recommended safety measures that can be taken to minimize risk and maximize benefit for patients in need of imaging. However, there are fewer data on performing MRIs in pacemaker-dependent patients with ICDs, who were excluded from the largest published study as well as the MagnaSafe Registry. Thus, demonstrating the safety and clinical utility of performing MRIs in this context is of high importance.

In response to urgent clinical considerations, Beth Israel Deaconess Medical Center has established a clinical protocol to provide safe MRIs in cases of compelling clinical indications, with close supervision and oversight from Radiology and Cardiac Electrophysiology staff. Thus, the investigators now propose a prospective study to evaluate safety and clinical outcomes for patients treated under this clinical protocol.

Specifically, this study proposes to perform a prospective clinical trial in patients with CIEDs that have a clinical need for MRI as outpatients to determine:

1. Safety according to the incidence rates of acute major and minor adverse events according to pre-specified definitions.
2. Clinical outcomes and scan utility affecting patients' survival and quality of life and treatment, including acute and longitudinal changes in device parameters, the need for system revision, and proportion of MRI findings influencing clinical management including medical or surgical interventions, and diagnostic or prognostic changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients have a medically/clinically indicated need for an MRI
* Patients with a non-MRI conditional pacemaker and/or ICD implanted after the year 2000
* Patients are willing and able to sign consent and HIPAA authorization or an authorized representative of the patient is willing to sign consent for the patient

  *The following factors are considered relative contraindications to the clinical protocol at BIDMC, and will similarly be considered exclusion criteria for the study. Exceptions on a case-by-case basis for circumstances of dire, life-threatening need may be considered.
* Leads implanted <6 weeks prior to the MRI
* Presence of any capped/abandoned leads
* Presence of nontransvenous epicardial leads

Exclusion Criteria:

* Other contraindications to MRI (e.g. other non-MRI-conditional implants)
* Pacemaker or ICD implanted prior to the year 2000
* Leads and/or generator implanted within 6 weeks of the proposed MRI
* CIED that is FDA approved as MRI conditional
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study of patients with a cardiac implantable electronic device (CIED) referred for a clinicially indicated MRI.
Sampling Method: Non-Probability Sample
Enrollment: 1169 (Actual)
Dates: Start 2016-12; Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Any of the Following Major Adverse Events | Change from baseline at 1 week and 6 months
  1. Acute loss of pacing peri-MRI (defined in scanner, or after scan prior to discharge)
  2. Inappropriate shock or ATP therapy peri-MRI
  3. Any death peri-MRI adjudicated to be related to the scan
Number of Patients with Any of the Following Minor Adverse Events | Change from baseline at 1 week and 6 months
  1. Clinically significant (symptoms or hemodynamic compromise) inappropriate pacing (e.g. undersensing or inappropriate asynchronous pacing)
  2. Any clinically significant arrhythmias peri-MRI
  3. Power-on-reset events
  4. Acute variation in pre/post MRI capture thresholds ≥ 50%
  5. Acute variation in pre/post MRI lead impedance ≥ 30%
  6. Acute variation in pre/post MRI P/R wave amplitude ≥ 50%

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kramer, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nazarian S, Reynolds MR, Ryan MP, Wolff SD, Mollenkopf SA, Turakhia MP. Utilization and likelihood of radiologic diagnostic imaging in patients with implantable cardiac defibrillators. J Magn Reson Imaging. 2016 Jan;43(1):115-27. doi: 10.1002/jmri.24971. Epub 2015 Jun 27. PMID 26118943
- [Background] Smith-Bindman R, Miglioretti DL, Larson EB. Rising use of diagnostic medical imaging in a large integrated health system. Health Aff (Millwood). 2008 Nov-Dec;27(6):1491-502. doi: 10.1377/hlthaff.27.6.1491. PMID 18997204
- [Background] Naehle CP, Strach K, Thomas D, Meyer C, Linhart M, Bitaraf S, Litt H, Schwab JO, Schild H, Sommer T. Magnetic resonance imaging at 1.5-T in patients with implantable cardioverter-defibrillators. J Am Coll Cardiol. 2009 Aug 4;54(6):549-55. doi: 10.1016/j.jacc.2009.04.050. PMID 19643318
- [Background] Naehle CP, Meyer C, Thomas D, Remerie S, Krautmacher C, Litt H, Luechinger R, Fimmers R, Schild H, Sommer T. Safety of brain 3-T MR imaging with transmit-receive head coil in patients with cardiac pacemakers: pilot prospective study with 51 examinations. Radiology. 2008 Dec;249(3):991-1001. doi: 10.1148/radiol.2493072195. PMID 19011193
- [Background] Sommer T, Naehle CP, Yang A, Zeijlemaker V, Hackenbroch M, Schmiedel A, Meyer C, Strach K, Skowasch D, Vahlhaus C, Litt H, Schild H. Strategy for safe performance of extrathoracic magnetic resonance imaging at 1.5 tesla in the presence of cardiac pacemakers in non-pacemaker-dependent patients: a prospective study with 115 examinations. Circulation. 2006 Sep 19;114(12):1285-92. doi: 10.1161/CIRCULATIONAHA.105.597013. Epub 2006 Sep 11. PMID 16966587
- [Background] Nazarian S, Hansford R, Roguin A, Goldsher D, Zviman MM, Lardo AC, Caffo BS, Frick KD, Kraut MA, Kamel IR, Calkins H, Berger RD, Bluemke DA, Halperin HR. A prospective evaluation of a protocol for magnetic resonance imaging of patients with implanted cardiac devices. Ann Intern Med. 2011 Oct 4;155(7):415-24. doi: 10.7326/0003-4819-155-7-201110040-00004. PMID 21969340
- [Background] Expert Panel on MR Safety; Kanal E, Barkovich AJ, Bell C, Borgstede JP, Bradley WG Jr, Froelich JW, Gimbel JR, Gosbee JW, Kuhni-Kaminski E, Larson PA, Lester JW Jr, Nyenhuis J, Schaefer DJ, Sebek EA, Weinreb J, Wilkoff BL, Woods TO, Lucey L, Hernandez D. ACR guidance document on MR safe practices: 2013. J Magn Reson Imaging. 2013 Mar;37(3):501-30. doi: 10.1002/jmri.24011. Epub 2013 Jan 23. PMID 23345200
- [Background] Levine GN, Gomes AS, Arai AE, Bluemke DA, Flamm SD, Kanal E, Manning WJ, Martin ET, Smith JM, Wilke N, Shellock FS; American Heart Association Committee on Diagnostic and Interventional Cardiac Catheterization; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Cardiovascular Radiology and Intervention. Safety of magnetic resonance imaging in patients with cardiovascular devices: an American Heart Association scientific statement from the Committee on Diagnostic and Interventional Cardiac Catheterization, Council on Clinical Cardiology, and the Council on Cardiovascular Radiology and Intervention: endorsed by the American College of Cardiology Foundation, the North American Society for Cardiac Imaging, and the Society for Cardiovascular Magnetic Resonance. Circulation. 2007 Dec 11;116(24):2878-91. doi: 10.1161/CIRCULATIONAHA.107.187256. Epub 2007 Nov 19. PMID 18025533
- [Background] Russo RJ. Determining the risks of clinically indicated nonthoracic magnetic resonance imaging at 1.5 T for patients with pacemakers and implantable cardioverter-defibrillators: rationale and design of the MagnaSafe Registry. Am Heart J. 2013 Mar;165(3):266-72. doi: 10.1016/j.ahj.2012.12.004. Epub 2013 Jan 28. PMID 23453091
- [Background] Cohen JD, Costa HS, Russo RJ. Determining the risks of magnetic resonance imaging at 1.5 tesla for patients with pacemakers and implantable cardioverter defibrillators. Am J Cardiol. 2012 Dec 1;110(11):1631-6. doi: 10.1016/j.amjcard.2012.07.030. Epub 2012 Aug 23. PMID 22921995